CLINICAL TRIAL: NCT06808217
Title: A Registry on the FARAVIEW Technology of the OPAL HDx Mapping System When Used With the FARAWAVE NAV Ablation Catheter in the Treatment of Atrial Fibrillation
Acronym: OPALISE
Status: Recruiting | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: PF337
Record Dates: First submitted 2025-01-29; First posted 2025-02-05 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation; Pulsed Field Ablation; FARAPULSE
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: FARAPULSE Pulsed Field Ablation System — Subjects who have provided written informed consent are considered enrolled. Subjects who have received ablation treatment with the FARAPULSE™ System are assigned to the 'TREATMENT' group.

SUMMARY:
The study is designed to collect data on the acute and long-term (1 year) safety and effectiveness outcome when an ablation procedure is performed in a commercial and standard of care setting with the FARAPULSE™ Pulsed Field Ablation System, whereby the FARAWAVE NAV Ablation catheter is used in conjunction with the OPAL HDx Mapping System. In addition, the study intends to analyse the association between several workflow-related variables, inclusive of intracardiac electro-anatomical mapping and ablation strategy with procedure-related complications (safety parameters), and one-year effectiveness parameters.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are prospectively planned and intended to be treated with the FARAPULSE™ Pulsed Field Ablation system for cardiac tissue ablation, per physician's medical judgement, and as per hospitals' standard of care
* Subjects who are willing and capable of providing informed consent
* Subjects who are willing and capable of participating to this Registry at an approved clinical investigational center
* Subjects whose age is 18 years or above, or who are of legal age to give informed consent specific to state and national law
* Subjects are planned to undergo an ablation procedure whereby the FARAWAVE NAV PF Ablation Catheter is used in conjunction with the OPAL HDx Mapping System.

Exclusion Criteria:

* Subjects who are currently enrolled in another investigational study or registry that would directly interfere with the current study. Exceptions are when the subject is participating in a mandatory governmental registry, or a purely observational registry, that do not interfere with the current study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: • Subjects who will undergo an ablation procedure with the FARAPULSE™ Pulsed Field Ablation system, per physician's medical judgement, and according to hospitals' standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint | 12 months
  The Primary Safety Endpoint is defined as the rate of device or procedure related serious adverse events following the index procedure through the 12 Month Follow-up
Primary effectiveness Endpoint | 12 Months
  The Primary Effectiveness Endpoint is defined as the rate of treatment success, which is defined by Acute and Chronic Procedural Success

CONTACTS AND LOCATIONS:
Locations (31):
- Allgemeines Krankenhaus AKH, Vienna, Austria
- Klinicki bolnicki centar Zagreb, Zagreb, Croatia
- France (7):
  - CHRU de Clermont-Ferrand, Clermont-Ferrand
  - CHU Grenoble, Grenoble
  - Hospital de la Pitie-Salpetriere, Paris
  - Hospital Europeen Georges-Pompidou (HEGP), Paris
  - Centre Cardiologique du Nord, Saint-Denis
  - CHU de Saint-Etienne, Saint-Priest-en-Jarez
  - Clinique Pasteur, Toulouse
- Germany (3):
  - Vivantes Klinikum Am Urban, Berlin
  - MVZ CCB Frankfurt und Main-Taunus GbR, Frankfurt
  - Asklepios Klinik Saint Georg, Hamburg
- Greece (2):
  - Henry Dunant Hospital Center, Athens
  - Ippokrateio General Hospital, Thessaloniki
- Mater Private Hospital, Dublin, Ireland
- Italy (3):
  - Maria Cecilia Hospital, Cotignola
  - Clinica Montevergine, Mercogliano
  - Ospedale Civile Di Piacenza, Piacenza
- Sheikh Jaber Al Ahmad Hospital, Kuwait City, Kuwait
- Centre Hospitalier Princesse Grace, Monaco, Monaco
- Netherlands (2):
  - Eramus MC- University Medical Center, Rotterdam
  - Isala Klinieken, Zwolle
- Poland (2):
  - Uniwersyteckie Centrum Kliniczne Warszawskiego Uniwersytetu Medycznego, Warsaw
  - Uniwersytecki Szpital Kliniczny Wrocławiu, Wroclaw
- National Guard Hospital, Riyadh, Saudi Arabia
- Spain (3):
  - Hospital de Basurto, Bilbao
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Marques de Valdecilla, Santander
- Switzerland (2):
  - Cardiocentro Ticino, Lugano
  - University Hospital Zurich, Zurich
- Cleveland Clinic London, London, United Kingdom